CLINICAL TRIAL: NCT04388787
Title: Investigating the Effect of Stochastic Resonance Vibration on Gait and Balance and Upper Extremity Function in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HM20018459
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- stochastic resonance (SR) vibration (Experimental): SR applied sub threshold at 90% of participant's detection threshold
  Interventions: Device: Stochastic resonance (SR) wraps
- Sham treatment (Sham Comparator): SR devices worn but not turned on (0% of participant's detection threshold).
  Interventions: Device: Stochastic resonance (SR) wraps
- Unblinded treatment (Experimental): SR is applied above participant's detection threshold at a participant selected intensity.
  Interventions: Device: Stochastic resonance (SR) wraps

INTERVENTIONS:
Device: Stochastic resonance (SR) wraps — SR wraps will be applied to the one or both wrists depending on whether the impairment is unilateral or bilateral. Two additional actuators will be secured around the shoulder. The threshold for detection of SR will be determined by the examiner prior to initiating the test condition. The intensity of the stimulation is adjustable with a scroll bar on the app and ranges from a 0 - 100. The examiner will gradually increase the stimulus intensity until the participant reports being able to feel it. This will set the participant's detection threshold.

SUMMARY:
The purpose of this research study is to determine the effects of wearable vibration devices for children with cerebral palsy and impaired arm function.

DETAILED DESCRIPTION:
Vibration devices have been used by some patients with cerebral palsy during therapy sessions. Researchers believe they have the potential to be even more useful for everyday use, and are doing this study to learn more about what they can do.

Participate in this study will be asked to complete assessments that test arm motion, muscle tone, motor control, and sensory function. They will then be asked to wear a wristband on each wrist and on their shoulder. These wristbands contain vibrators that can vibrate at different levels. The vibrations are caused by a low-level of sound waves that people may barely be able to hear. While wearing the vibration devices on the wrist and shoulder, participants will be asked to perform two tasks. The first task is called the box and blocks test, which consists of transferring wooden blocks from one box to another. The second test is called the Shriners upper extremity evaluation (SHUEE). In this test participants will perform a series of fine motor tasks with their hands. The SHUEE test will be video recorded for scoring by a study therapist at a later time on how much and how well participants use their impaired arm to perform the tasks. Participants will be asked to complete the box and blocks test and the SHUEE test 3 times. Participation in this study will be one single visit and last approximately an hour to an hour and a half.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy
* 3 years to 18 years of age
* Able to reliably express pain, discomfort or fear as reported by the parent/guardian
* Manual ability classification scale (MACS) levels I, II or III

Exclusion Criteria:

* Any unstable medical condition. An unstable medical condition is a state of imminent threat to life such as shock, acute asthma, respiratory distress, severe infection and sepsis. Any patient in a clinic or therapy center presenting with signs and symptoms of an unstable medical condition will be directed to emergency medical services
* Any medical condition preventing active rehabilitation reported by the parent/guardian such as:

  o Thromboembolic disease, acute progressive neurological disorder, cardiovascular or pulmonary contraindications, aggressive behavior, severe cognitive deficits, joint instabilities and compromised bone health, recent or non-consolidated fractures, osteoporosis
* Subjects with cardiac pacemakers, electronic pumps or any other implanted medical devices
* Skin lesions affecting the areas where the device straps will be attached to the body

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subthreshold, Sham, and Above Threshold Stochastic Resonance (SR) Vibration: There was only one arm to the study. Participants were not assigned to different arms based on order of treatment because treatment order was not relevant to the outcome and was not tracked in the data set. Each participant completed all treatments in one session. Order of blinded and sham treatments was randomized at the time data was collected. The unblinded treatment was always last.
  Stochastic resonance (SR) wraps: SR wraps were applied to the one or both wrists depending on whether the impairment is unilateral or bilateral. Two additional actuators were secured around the shoulder. The threshold for detection of SR was determined by the examiner prior to initiating the test condition. The intensity of the stimulation was adjustable with a scroll bar on the app and ranged from a 0 - 100. The examiner gradually increased the stimulus intensity until the participant reported being able to feel it. This set the participant's detection threshold.
  Once the detection threshold was established, participant completed the assessments under 3 treatments, the first two in random order and the third always last:
  Blinded: SR applied sub threshold at 90% of participant's detection threshold
  Blinded Sham: SR devices worn but not turned on (0% of participant's detection threshold).
  Unblinded: SR is applied above participant's detection threshold at a participant selected intensity.
Period: Blinded Period
Arm/Group | Subthreshold, Sham, and Above Threshold Stochastic Resonance (SR) Vibration
Started | 16
Completed First Assessment - Approximately 15 Minutes (Specific Treatment Unknown) | 15
Completed Second Assessment - Approximately 15 Minutes (Specific Treatment Unknown) | 15
Completed | 15
Not Completed | 1
Not completed — Patient could not follow instructions | 1
Period: Unblinded Period
Arm/Group | Subthreshold, Sham, and Above Threshold Stochastic Resonance (SR) Vibration
Started | 15
Completed | 6
Not Completed | 9
Not completed — Patients became fatiged after a single round of testing with sham vs subthreshold | 9

BASELINE CHARACTERISTICS:
Arm/Group | Subthreshold, Sham, and Above Threshold Stochastic Resonance (SR) Vibration
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Manual Dexterity
Description: Manual dexterity is will be assessed using the Box and Block (B&B) test. The B&B test is scored by counting the number of blocks transferred during the 1 minute test. Higher scores indicate better manual dexterity. Change was assessed after each condition and compared to baseline.
Time Frame: Baseline to up to 1.5 hours
Population: Data from all participants who completed the blinded portion of the study were analyzed for the subthreshold and sham treatments. Only participants who completed the unblinded portion were analyzed for the above threshold treatment
Measure: Mean (Standard Deviation); unit: points on assessment
Groups:
- Blinded Subthreshold Stochastic Resonance (SR) Vibration: Stochastic resonance (SR) wraps: SR wraps were applied to the one or both wrists depending on whether the impairment is unilateral or bilateral. Two additional actuators were secured around the shoulder. The threshold for detection of SR was determined by the examiner prior to initiating the test condition. The intensity of the stimulation was adjustable with a scroll bar on the app and ranged from a 0 - 100. The examiner gradually increased the stimulus intensity until the participant reported being able to feel it. This set the participant's detection threshold.
  Once the detection threshold was established, participant completed the assessments with SR vibration applied sub threshold at 90% of participant's detection threshold.
- Blinded Sham Treatment: Stochastic resonance (SR) wraps: SR wraps were applied to the one or both wrists depending on whether the impairment is unilateral or bilateral. Two additional actuators were secured around the shoulder. The threshold for detection of SR was determined by the examiner prior to initiating the test condition. The intensity of the stimulation was adjustable with a scroll bar on the app and ranged from a 0 - 100. The examiner gradually increased the stimulus intensity until the participant reported being able to feel it. This set the participant's detection threshold.
  Once the detection threshold was established, participant completed the assessments with SR devices worn but not turned on (0% of participant's detection threshold).
- Unblinded Above Threshold SR Vibration: Stochastic resonance (SR) wraps: SR wraps were applied to the one or both wrists depending on whether the impairment is unilateral or bilateral. Two additional actuators were secured around the shoulder. The threshold for detection of SR was determined by the examiner prior to initiating the test condition. The intensity of the stimulation was adjustable with a scroll bar on the app and ranged from a 0 - 100. The examiner gradually increased the stimulus intensity until the participant reported being able to feel it. This set the participant's detection threshold.
  Once the detection threshold was established, participant completed the assessments SR is applied above participant's detection threshold at a participant selected intensity.
Arm/Group | Blinded Subthreshold Stochastic Resonance (SR) Vibration | Blinded Sham Treatment | Unblinded Above Threshold SR Vibration
Number analyzed (Participants) | 15 | 15 | 6
points on assessment | 10.7 (7.1) | 12.4 (6.4) | 14.4 (6.7)
Statistical Analysis 1: Comparison: Blinded Subthreshold Stochastic Resonance (SR) Vibration vs Blinded Sham Treatment vs Unblinded Above Threshold SR Vibration; Test type: Superiority; p = 0.03, ANCOVA

2. Primary Outcome: Change in Upper Extremity Functionality
Description: Upper extremity functionality will be assessed using the Shriners Upper Extremity Evaluation (SHUEE). Participants are observed and scored by a trained rater blind to the condition. Scores range from 0 to 45 for spontaneous functional activity and from 0 to 72 for dynamic positional analysis. Higher scores indicate better functionality.
Time Frame: Baseline to up to 1.5 hours
Measure: Mean (Standard Deviation); unit: points on assessment
Arm/Group | Blinded Subthreshold Stochastic Resonance (SR) Vibration | Blinded Sham Treatment | Unblinded Above Threshold SR Vibration
Number analyzed (Participants) | 15 | 15 | 6
points on assessment
  spontaneous functional analysis | 21.2 (4.9) | 24.2 (8.8) | 30.8 (4.9)
  dynamic positional analysis | 37.1 (13.1) | 34.4 (10.0) | 48.6 (12.2)
Statistical Analysis 1: Comparison: Blinded Subthreshold Stochastic Resonance (SR) Vibration vs Blinded Sham Treatment vs Unblinded Above Threshold SR Vibration; Test type: Superiority; p = 0.0008, ANCOVA

ADVERSE EVENTS:
Time Frame: 90 minutes
Arm/Group | Blinded Subthreshold Stochastic Resonance (SR) Vibration | Blinded Sham Treatment | Unblinded Above Threshold SR Vibration
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/6
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04388787/Prot_SAP_000.pdf